CLINICAL TRIAL: NCT05619263
Title: Emergency Preparedness and Support for Caregivers of Persons With Dementia: Disaster PrepWise
Brief Title: Emergency Preparedness for Caregivers of Persons With Dementia: Disaster PrepWise
Acronym: DPW-Caregiver
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sato Ashida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Sato Ashida, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 202201195; 1R01AG077436 (NIH)
Record Dates: First submitted 2022-11-02; First posted 2022-11-16 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-06

CONDITIONS: Caregiver Resilience and Stress
Keywords: Alzheimer's disease; Dementia; Caregiver; Disaster preparedness
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Caregivers who consent to participate, complete a baseline survey, and are assigned to the control arm will receive a four-page handout on Emergency Preparedness published by the Alzheimer's Association that provides tips on preparing for disasters and what to do during and after a disaster. Control participants will complete follow-up surveys at 3 and 6 months, similar to intervention participants.
- Disaster PrepWise-Caregiver Intervention (Experimental): Caregivers who consent to participate, complete a baseline survey, and are assigned to the intervention arm will receive a Disaster PrepWise-Caregiver program from a trained interventionist and receive a completed household emergency management plan. Control participants will complete follow-up surveys at 3 and 6 months, similar to intervention participants.
  Interventions: Behavioral: Disaster PrepWise-Caregiver

INTERVENTIONS:
Behavioral: Disaster PrepWise-Caregiver — The Disaster PrepWise (DPW) intervention consists of five interactive modules and two supplemental sections (special topics and resources on various types of disasters). The five modules are: (1) Complete a Personal & Household Assessment, (2) Develop a Personal Emergency Network, (3) Develop Emergency Information & Gather Important Documents, (4) Keep a 3-5 Day Supply of Medications & Medical Supplies, and (5) Build an Emergency Supply Kit. Through an initial visit (IV1) and a follow-up phone conversation 4 weeks later (IV2), the interventionist will develop a personalized disaster management plan and provide it to the participant for sharing with family and friends. Eight weeks after the initial session, the interventionist will make a final follow-up call (IV3) to provide any additional assistance caregivers may need.
  Arms: Disaster PrepWise-Caregiver Intervention

SUMMARY:
Individuals with dementia and their families are especially vulnerable during a disaster as it limits caregivers' ability to continue with care due to disaster related stress and reduced access to resources and support. The COVID-19 pandemic showed the extreme vulnerability of persons with dementia (PWD) and their caregivers as they struggled to access support and resources due to the threat of COVID-19 infection; such impact was exacerbated in rural areas where caregivers are geographically isolated and disaster management resources are scarce. With the number of federally declared disasters increasing dramatically over the past 50 years, active public health efforts are needed to support caregivers in developing emergency caregiving plans usable in disasters such as pandemics and extreme weather emergencies. The long-term goal of this project is to enhance emergency preparedness and support networks of caregivers of PWD to increase their resilience and minimize distress by implementing an intervention program, Disaster PrepWise (DPW). In the DPW program, a trained Medical Reserve Corp (MRC) volunteer will provide step-by-step guidance to caregivers to jointly develop emergency preparedness plans and personal support networks. The objectives of this proposed study are to 1) test the impact of DPW on caregiver outcomes (i.e., resilience, stress) and perceptions that may mediate the association between DPW and outcomes (caregiver self-efficacy, preparedness, social support); and 2) evaluate implementation strategies in a real-world setting to optimize future dissemination. We will conduct a randomized control trial of 250 caregivers of persons with dementia involving two arms: DPW intervention group and an information-only control group (print information on disaster preparedness). Assessments will occur before randomization (baseline), and 3 and 6 months after the baseline. This study is innovative in its use of a highly personalized disaster preparedness program with built-in assistance to support caregivers; the support will be provided through an existing national-level public health infrastructure (MRC) that has a great potential to reach older adults and caregivers in rural areas. The knowledge and data obtained through this study will lay the foundation for a future larger-scale multi-state pragmatic trial to assess dissemination potentials.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adults (18 years and older)
* Family members (e.g., biological and non-biological relatives, friends) of individuals diagnosed with ADRD regardless of whether they live with the individual or not. Individuals will not be excluded based on race/ethnicity, gender, or sexual orientation.

Exclusion Criteria:

* Families of those diagnosed as predementia or mild cognitive impairment are excluded from the parent study due to differing care needs.
* DPW addresses the needs of community-dwelling individuals, thus, caregivers of those living in nursing homes facilities will be excluded.
* Caregivers with physical or cognitive conditions that prevent them from consenting or providing responses to questions will be excluded following evaluation ("Evaluation to Sign an Informed Consent Document for Research," UI IRB).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Resilience | Change between baseline and 6-month follow-up
  Connor-Davidson Resilience Scale (CD-RISC: 25 items). The range is 0 to 100. Higher scores indicate higher resilience.
Caregiver stress | Change between baseline and 6-month follow-up
  Cohen Perceived Stress Scale (PSS: 14 items). The range is 0 to 40. Higher scores indicate higher perceived stress.

SECONDARY OUTCOMES:
Self-Efficacy | Change between baseline and 6-month follow-up
  Caregiver Self-Efficacy (SE to manage care, 5 items; SE to use services, 4 items). The range is 0-10. A higher score indicates a higher amount of self-efficacy.
Caregiver Preparedness | Change between baseline and 6-month follow-up
  Caregiver Preparedness scale (8 items). The range is 0 to 40. A higher score indicates that the caregiver feels more prepared for caregiving.
Social Networks | Change between baseline and 6-month follow-up
  CaREnet: Caregiver Social Network Assessment tool. It is not a scale score. Counts of network members engaging in supportive interactions.

CONTACTS AND LOCATIONS:
Overall Officials: Sato Ashida, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No